CLINICAL TRIAL: NCT00999089
Title: Arrested Versus Beating Heart Techniques in Coronary Revascularisation: Randomized Clinical Trial in Unselected Patients
Brief Title: Arrested Versus Beating Heart Techniques in Coronary Revascularisation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Jochen Boergermann, Martin-Luther-University Halle-Wittenberg, Department of Cardiothoracic Surgery
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3CAB-STUDY
Record Dates: First submitted 2009-10-19; First posted 2009-10-21 (Estimated); Last update posted 2009-10-21 (Estimated); Status verified 2009-10

CONDITIONS: Coronary Artery Bypass Grafting
Keywords: Coronary disease; Coronary artery bypass grafting; Cardiopulmonary bypass; Extracorporeal circulation; Cardioplegia; Off pump
MeSH Terms: conditions — Coronary Disease | interventions — Coronary Artery Bypass, Off-Pump

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- CCAB (Active Comparator): Conventional Coronary Artery Bypass
  Interventions: Procedure: Conventional Coronary Artery Bypass
- OPCAB (Active Comparator): Off-Pump Coronary Artery Bypass
  Interventions: Procedure: Off-Pump Coronary Artery Bypass
- PACAB (Active Comparator): Pump-Assisted Coronary Artery Bypass
  Interventions: Procedure: Pump-Assisted Coronary Artery Bypass

INTERVENTIONS:
Procedure: Conventional Coronary Artery Bypass — Coronary artery bypass grafting with extracorporeal circulation and cardioplegic arrest
  Arms: CCAB
Procedure: Off-Pump Coronary Artery Bypass — Coronary artery bypass grafting without extracorporeal circulation or global myocardial ischemia
  Arms: OPCAB
Procedure: Pump-Assisted Coronary Artery Bypass — Coronary artery bypass grafting with a beating but unloaded heart by using extracorporeal circulation
  Arms: PACAB

SUMMARY:
The individual contribution of the specific injuring mechanisms surgical trauma, extracorporeal circulation, and ischemia/reperfusion to clinical outcome in coronary revascularisation remains to be elucidated. The effect of these factors is analyzed in this randomized clinical trial by comparing the 3 surgical approaches: Conventional Coronary Artery Bypass Grafting (CCAB), with extracorporeal circulation and cardioplegic arrest; Off-Pump Coronary Artery Bypass Grafting (OPCAB), avoids extracorporeal circulation and global myocardial ischemia; and Pump-Assisted Coronary Artery Bypass Grafting (PACAB), with an unloaded and beating heart. The hypothesis addressed by the study is that the surgical invasiveness increases in the order: OPCAB, PACAB, CCAB.

ELIGIBILITY:
Inclusion Criteria:

* patients with double- or triple-vessel coronary artery disease
* patients with left ventricular ejection fraction =< 40% or >= 60%
* elective or urgent isolated coronary artery bypass grafting

Exclusion Criteria:

* previous cardiac surgery
* emergency indications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 616 (Actual)
Dates: Start 2003-01; Primary Completion 2006-09 (Actual); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
All cause mortality | 1, 6, 12, 24, 48 month
Myocardial infarction | 1, 6, 12, 24, 48 month
Stroke | 1, 6, 12, 24, 48 month
Low-output syndrome | in hospital
duration of ventilation >= 24h | in hospital
New requirement of hemodialysis | in hospital

SECONDARY OUTCOMES:
Completeness of revascularization | in hospital
Re-revascularization of the target vessel (PCI and/or CABG) | 1, 6, 12, 24, 48 month
Resource use (operative time, duration of stay in the intensive care unit, total hospital stay) | in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Boergermann, MD, Principal Investigator — Martin-Luther-University Halle-Wittenberg; Rolf E Silber, MD, Study Chair — Martin-Luther-University Halle-Wittenberg
Locations (2):
- Germany (2):
  - Heart Center Coswig, Department of Cardiothoracic and Vascular Surgery, Coswig
  - Martin-Luther-University Halle-Wittenberg, Department of Cardiothoracic Surgery, Halle